CLINICAL TRIAL: NCT02120547
Title: An Open Label, Phase 1 Study to Evaluate the Effect of Mile and Moderate Hepatic Impairment on the Multiple-Dose Pharmacokinetics of Cenicriviroc (CVC)
Brief Title: Phase 1 Study of Multiple-Dose Pharmacokinetics of Cenicriviroc in Subjects With Mild and Moderate Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: TBR 652-1-121
Record Dates: First submitted 2014-04-18; First posted 2014-04-22 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Liver Insufficiency
Keywords: Liver Insufficiency; Hepatic impairment
MeSH Terms: conditions — Hepatic Insufficiency | interventions — cenicriviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cenicriviroc in mild liver impaired (Experimental): Subjects with mild liver impaired will receive cenicriviroc, 1 tablet once daily, for 14 days. Matching healthy subjects will receive Cenicriviroc, 1 tablet once daily, for 14 days.
  Interventions: Drug: Cenicriviroc in mild liver impaired
- Cenicriviroc in moderate liver impaired (Experimental): Subjects with moderate liver impaired will receive cenicriviroc, 1 tablet once daily, for 14 days. Matching healthy subjects will receive Cenicriviroc, 1 tablet once daily, for 14 days.
  Interventions: Drug: Cenicriviroc in moderate liver impaired

INTERVENTIONS:
Drug: Cenicriviroc in mild liver impaired — Subjects with mild hepatic impairment will receive CVC, 1 tablet once daily, for 14 days. Matching healthy subjects will receive CVC, 1 tablet once daily, for 14 days.
  Other Names: CVC
  Arms: Cenicriviroc in mild liver impaired
Drug: Cenicriviroc in moderate liver impaired — Subjects with moderate hepatic impairment will receive CVC, 1 tablet once daily, for 14 days. Matching healthy subjects will receive CVC, 1 tablet once daily, for 14 days.
  Other Names: CVC
  Arms: Cenicriviroc in moderate liver impaired

SUMMARY:
To determine whether CVC exposures are altered in subjects with impaired hepatic function, compared to subjects with normal hepatic function. The results will help guide the clinical use of CVC in patients with hepatic impairment, determine the extent of PK changes, if any, and identify the potential need for dose adjustments of CVC in this population.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females aged 18-65
* Weight ≥ 50.0 kg
* BMI 18.0 - 40.0 kg/m2
* Able to participate, and willing to give written informed consent and to comply with the study restrictions
* Subjects with hepatic impairment will have stable liver disease (Child Pugh A or Child Pugh B)

Exclusion Criteria:

* Pregnant or lactating women and male partners of women who are pregnant or lactating
* Uncontrolled treated or untreated hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 105 mmHg)
* QTcF > 450 msec for males and > 470 msec for females at Screening or Day -1
* Donation or loss of blood over 350 mL within 60 days prior to screening
* Any evidence of progressive liver disease within the last 4 weeks for subjects with hepatic impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Multiple-dose pharmacokinetics of CVC | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12 and 24 hours postdose on Days 1 and 14
  Intensive PK on Days 1 and 14. Trough PK on Days 3-13. Additional free (unbound) CVC will be assessed 2 hours and 24 hours postdose on Day 14.

SECONDARY OUTCOMES:
Safety and tolerability | Days 1 through 35 for hepatic impaired subjects and Days 1-28 for healthy matching subjects
  Adverse events, concomitant medications, vital signs, 12-lead triplicate ECGs, clinical laboratory tests (chemistry, hematology, urinalysis) and physical examinations will be assessed.

OTHER OUTCOMES:
Pro-inflammatory cytokines and biomarkers of bacterial translocation | 28 days after receiving first dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth C Lasseter, MD, Principal Investigator — Clinical Pharmacology of Miami, Inc.
Locations (1):
- Clinical Pharmacology of Miami, Inc., Fort Lauderdale, Florida, United States